CLINICAL TRIAL: NCT05324293
Title: An Open Label Study, to Evaluate Safety, Tolerability, and Efficacy in Male and Female with Androgenetic Alopecia Treated with HMI-115 Over a 24-Week Treatment Period
Brief Title: To Evaluate the Safety, Tolerability and Efficacy in Male and Female with AGA Treated with HMI-115 Over a 24-week Treatment Period
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hope Medicine (Nanjing) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMI-115102
Record Dates: First submitted 2022-03-30; First posted 2022-04-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-10

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HMI-115 240mg (Experimental)
  Interventions: Drug: HMI-115

INTERVENTIONS:
Drug: HMI-115 — Once Every 2 weeks, subcutaneously injection

SUMMARY:
An Open Label Study, to Evaluate Safety, Tolerability, and Efficacy Study in Male and Female with Androgenetic Alopecia Treated with HMI-115 over a 24-Week Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Male and Female subjects, between 18 and 65 years of , inclusive, at the time of signing informed consent.
3. Clinical diagnosis of androgenetic alopecia. Male subjects who meet Norwood-Hamilton scales 3v, 4 and 5. Female subjects who meet Sinclair scales 2-4.

Exclusion Criteria:

1. Subject with clinical diagnosis of non-AGA
2. Subject with clinically relevant abnormal skin or scalp findings which could interfere study assessment
3. Subject has used therapies associated with hair growth or may affect PRL levels, within defined time window before Screening
4. Subject with history of anterior pituitary, posterior pituitary, or hypothalamic dysfunction
5. Subject has clinically significantly abnormal laboratory tests at Screening
6. Known hypersensitivity to any of the IMP ingredients
7. Any other conditions in the investigator's opinion that prevent the subject from participating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
TAHC(target area hair count) of non-vellus | From baseline to Week 24
  Change in target area hair count (TAHC) of non-vellus from baseline to Week 24 in male and female AGA subjects, respectively.

SECONDARY OUTCOMES:
TAHC of non-vellus | From baseline to Week 6, 12, 18, and 36
  Change in TAHC of non-vellus from baseline to Week 6, 12, 18, and 36 in male and female, respectively.
TAHW(target area hair width) of non-vellus hair | From baseline to Week 6, 12, 18, 24, and 36
  Change in target area hair width (TAHW) of non-vellus hair from baseline to Week 6, 12, 18, 24, and 36 in male and female, respectively.
Investigator Global Assessment (IGA) | Week 6, 12, 18, 24, and 36
  IGA at Week 6, 12, 18, 24, and 36 in male and female, respectively.
Subject self-Assessment (SSA) | Week 6, 12, 18, 24, and 36
  SSA at Week 6, 12, 18, 24, and 36 in male and female, respectively.
Hair growth questionnaire assessment (HGQA) | Week 6, 12, 18, 24, and 36
  HGQA at Week 6, 12, 18, 24, and 36 in male and female, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Rodney Sinclair Pty Ltd, trading as Sinclair Dermatology, Melbourne E., Victoria, Australia